CLINICAL TRIAL: NCT02357212
Title: Early Invasive Versus Conservative Therapy in Women With an Acute Coronary Syndrome
Acronym: Lady Gator
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00-2008
Record Dates: First submitted 2015-01-23; First posted 2015-02-06 (Estimated); Last update posted 2015-02-16 (Estimated); Status verified 2015-02

CONDITIONS: Acute Coronary Syndrome
Keywords: Non-St elevation acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Exercise Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Invasive (Other): Patients assigned to an early invasive strategy will undergo coronary angiography within 48 hours and have percutaneous coronary intervention or coronary artery bypass grafting performed as soon as possible during the initial hospitalization if deemed appropriate.
  Interventions: Procedure: coronary angiography
- Conservative management (Other): Patients assigned to conservative management will be treated with anti-anginal medications, aspirin, clopidogrel, atorvastatin, and other guideline recommended medicines. Patients will have an echocardiogram and adenosine stress testing
  Interventions: Procedure: adenosine stress test

INTERVENTIONS:
Procedure: coronary angiography — invasive procedure performed to determine coronary anatomy
  Arms: Early Invasive
Procedure: adenosine stress test — non-invasive procedure to determine area of cardiac ischemia
  Other Names: stress test
  Arms: Conservative management

SUMMARY:
The aim of this research is to evaluate the effect of early invasive therapy and appropriate revascularization compared with conservative management and selective revascularization among women with an acute coronary syndrome.

DETAILED DESCRIPTION:
This study aims to enroll 1,000 women who present with AcuteCoronarySyndorme ( ACS). Patients will be identified through screening of all women admitted for chest pain, and those women with positive cardiac enzymes after operative procedures. After receiving permission to approach the potential subjects, trained and delegated study personnel will present the study to the patient. The informed consent process will be completed by the study coordinator, PI or co-investigator. The patient will have all procedures, risks and benefits explained and offered time to read and review the informed consent form. They will be given adequate time to ask questions, consult with family members or primary physicians. Specifically, written informed consent will be obtained in the emergency department or in the cardiology ward/unit before the patient is sedated/in the catheterization laboratory. . When a patient consents to participate in the study, their treatment assignment will be randomly determined by opening a sealed envelope that contains one of two treatment strategies. The blinding envelopes will be created by the Biostatistics group and will be sealed.

Once informed written consent is obtained (see accompanying flow chart), each patient will be randomly assigned to early invasive therapy versus conservative management. All patients will be administered aspirin 325 mg, clopidogrel 600 mg, and atorvastatin 80 mg. Anti-thrombin therapy (unfractionated heparin or bivalirudin according to physician discretion) will be administered intravenously. If anti-thrombin therapy was administered prior to randomization, this agent will be continued through catheterization and titrated if necessary to achieve desired effect.

Patients assigned to an early invasive strategy will undergo coronary angiography within 48 hours and have percutaneous coronary intervention or coronary artery bypass grafting performed as soon as possible during the initial hospitalization if deemed appropriate. The choice of intervention or surgery will be determined by the operator according to coronary anatomy and consistent with current practice guidelines. For example, disease of the left main trunk, or multi-vessel disease would generally be expected to be referred for surgical revascularization. Patients who undergo percutaneous coronary intervention can receive a glycoprotein IIb/IIIa inhibitor (i.e. abciximab bolus by intra-coronary or intra-venous route (0.25 mg per kg), followed by infusion (0.125 µg per kg per minute for 12 hours). Upfront use of glycoprotein IIb/IIIa inhibitors is discouraged. Eptifibatide or tirofiban can be used instead of abciximab according to operator discretion. Elective percutaneous coronary intervention on non-culprit vessels, in either study arm, can take place sometime after the index procedure with the goal to achieve complete revascularization. Such staged procedures will not be adjudicated as an urgent need for revascularization.

Patients assigned to conservative management will be treated with anti-anginal medications, as well as aspirin, clopidogrel, atorvastatin, and other guideline recommended medicines. Anti-thrombin therapy will be continued for no more than 48 hours. Conservative therapy will continue during this time, unless the patient has refractory angina, hemodynamic or electrical instability, left ventricular dysfunction (left ventricular ejection fraction < 45%), or significant ischemia on predischarge stress testing. Patients will have an echocardiogram to determine left ventricle function. Stress testing will be performed by adenosine SPECT if there is no left ventricular dysfunction by echocardiography. Patients with any high risk findings, such as refractory chest pain, left ventricular ejection fraction < 45%, or a large burden of ischemia on stress testing will remain in the hospital to undergo cardiac catheterization.

Patients in both groups will be treated with lifelong aspirin, 12 months of clopidogrel, in addition to atorvastatin and other guideline recommended therapies. A shorter duration of clopidogrel can be recommended in select cases according to treating physician discretion.

Specific data for acquisition:

Protected health information will be accessed by the practitioners normally involved in the patient's care during their hospitalization. Research demographics will be obtained by the research coordinator by interviewing the patient and by chart review. After hospital discharge, the research coordinator will contact the patient at specified intervals to determine if an endpoint has been met. Evidence that an endpoint occurred would require additional supplemental chart review by the research coordinator.

Patient demographics: age, height, weight, body mass index, medications at randomization, pertinent medical/surgical/family/social history: for example hypertension, hypercholesterolemia, diabetes mellitus, current tobacco use, history of: prior myocardial infarction, percutaneous coronary intervention or coronary artery bypass grafting. This data will be gathered by the research coordinator through patient reporting and chart review.

Procedural: Duration of ischemic symptoms from onset until randomization, electrocardiographic changes, elevated cardiac biomarkers, elevated NT-pro-BNP, procedural success defined as Thrombolysis In Myocardial Infarction flow 3, drug-eluting stent use, glycoprotein IIb/IIIa inhibitor use, intra-procedural activated clotting time, closure device, sheath size, micropuncture access.

ELIGIBILITY:
Inclusion Criteria:

1. Women age 18 years or older
2. Non-ST-elevation acute coronary syndrome (defined as new onset chest discomfort that occurs at rest or with low levels of activity/or emotion within the preceding 48 hours) with either:

   1. elevated troponin T (≥ 0.03 ng per milliliter),
   2. elevated creatinine kinase MB-isoenzyme (≥ 5.0 ng per milliliter)
   3. elevated NT-pro-BNP (≥ 450 pg per milliliter),
   4. ST-segment depression (≥ 0.5 mm)
   5. or TIMI risk score (> 2)
3. women who have elevated cardiac enzymes after non-cardiac surgery will also be considered.

Exclusion Criteria:

1. ST-elevation myocardial infarction,
2. cardiogenic shock,
3. congestive heart failure,
4. hemodynamic instability,
5. use of fibrinolytic therapy in the last 96 hours,
6. current bleeding or bleeding disorder within the last 3 months that required transfusion,
7. pregnancy,
8. contraindication to any study medication. i.e.heparin, clopidogrel, or glycoprotein IIb/III inhibitor,
9. PCI in the last 6 months,
10. prior CABG,
11. inability to provide written informed consent.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
cumulative incidence of death | 1 year
  among women with an acute coronary syndrome between the 2 randomized treatment groups
cumulative incidence of myocardial infarction | 1 year
  among women with an acute coronary syndrome between the 2 randomized treatment groups
cumulative incidence of rehospitalization for ACS | 1 year
  among women with an acute coronary syndrome between the 2 randomized treatment groups
cumulative incidence of stroke | 1 year
  among women with an acute coronary syndrome between the 2 randomized treatment groups
cumulative incidence of major bleeding | 1 year
  among women with an acute coronary syndrome between the 2 randomized treatment groups

SECONDARY OUTCOMES:
Death | 6months, 1 year, 2 year
  Composite ischemic outcome
Myocardial Infarction | 6 months, 1 year, 2 year
  Composite ischemic outcome
Rehospitalization for ACS | 6 months, 1 year, 2 year
  Composite ischemic outcome
Stroke | 6 months, 1 year, 2 year
  Composite ischemic outcome
major bleeding | 6 months, 1 year, 2 year
  Composite ischemic outcome
Death | 6 months, 1 year, 2 year
  Individual components
Myocardial Infarction | 6 months, 1 year, 2 year
  Individual components
Stroke | 6 months, 1 year, 2year
  Individual components
Rehospitalization for ACS | 6 months, 1 year, 2 year
  Individual components
major bleeding | 6 months, 1 year, 2 year
  Individual components

OTHER OUTCOMES:
Urgent need for revascularization | 1 year
  percutaneous coronary intervention or coronary artery bypass grafting due to ischemic symptoms at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Anthony A Bavry, M.D., MPH, Principal Investigator — Universtiy of Florida